CLINICAL TRIAL: NCT01663103
Title: Interleukin-1 Trap to Treat Vascular Dysfunction in Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12-0586
Record Dates: First submitted 2012-08-07; First posted 2012-08-13 (Estimated); Results first posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Interleukin-1; Endothelium, Vascular; Vascular Stiffness; Oxidative Stress; Inflammation; Endothelial cells
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — rilonacept; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rilonacept (Experimental): 12 weeks of treatment with rilonacept
  Interventions: Drug: Rilonacept
- Placebo (Placebo Comparator): Twelve weeks of treatment with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilonacept — 12 weeks of treatment with rilonacept (subcutaneous injection with a loading dose of 320 mg, followed by 160 mg/wk)
  Other Names: Arcalyst
  Arms: Rilonacept
Drug: Placebo — Twelve weeks of treatment with placebo (subcutaneous injection of normal saline with a loading dose of 320 mg, followed by 160 mg/wk)
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
Risk of cardiovascular diseases (CVD) is significantly elevated in patients with chronic kidney disease (CKD); however, this increased risk is only partially explained by traditional cardiovascular risk factors. Patients with CKD exhibit chronic inflammation, a key mechanism contributing to vascular dysfunction (i.e., large elastic artery stiffening and endothelial dysfunction). Inhibiting inflammation improves vascular dysfunction in other populations characterized by chronic inflammation. However, it is currently unknown if reducing inflammation with an interleukin-1 (IL-1) blocker enhances vascular function in CKD patients. Aim 1 will assess the efficacy of IL-1 blocking with rilonacept for treating vascular dysfunction in patients with stage III or IV CKD (estimated glomerular filtration rate 15-60 mL/min/1.73 m2). Aim 2 will determine if blocking IL-1 with rilonacept also reduces inflammation and oxidative stress. These studies could shift clinical practice guidelines by establishing a novel therapy for reducing CVD risk in CKD patients not requiring chronic hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* CKD stage III or IV (eGFR with the 4-variable Modified Diet Renal Disease (MDRD) prediction equation: 15-60 mL/min/1.73m2; stable renal function in the past 3 months)
* An elevated high sensitivity C-reactive protein (hs-CRP) of > 2.0 mg/L and <30 mg/L on at least 2 consecutive weekly determinations
* Urine protein excretion < 5.0 g/24h estimated by a spot urine protein/creatinine ratio
* Ability to provide informed consent

Exclusion Criteria:

* Patients with advanced CKD requiring chronic dialysis
* Active infection (chronic or acute (within 3 months) or antibiotic therapy (w/in 1 mo); history of recurrent infection
* Significant co-morbid conditions that lead the investigator to conclude that life expectancy is less than 1 year
* Expected to undergo living related transplant in next 6 months
* History of severe congestive heart failure (i.e., EF < 35%)
* Hospitalization in the past month
* Severe arthritis, lupus, inflammatory bowel disease, asthma or other disease(s) or medical condition(s) that, in the opinion of the investigator, could interfere with hsCRP or immune function
* Immunosuppressant agents such as cyclosporine, tacrolimus, azathioprine, etanercept, infliximab, adalimumab, anakinra or long-term oral glucocorticoids taken in past 12 months
* Known malignancy
* HIV, active, chronic hepatitis B as evidenced by HBsAg positive and HBsAb negative, or hepatitis C positive
* Woman who are pregnant, nursing or planning to become pregnant
* Body mass index (BMI) >40 kg/m2
* Warfarin use (or other cytochrome P (CYP)450 substrates with a narrow therapeutic index) [ok if do not participate in endothelial cell collection]
* Taking medication(s) that interact with agents administered during experimental sessions (e.g., sildenafil interacts with nitroglycerin)
* Currently receiving or planning to receive live or inactivated vaccines
* Alcohol dependence or abuse
* Subjects at risk for tuberculosis (TB). Specifically, subjects with:
* Current clinical, radiographic or laboratory evidence of active TB at screening or latent TB that has not been previously treated
* A history of active TB within the last 3 years even if it was treated.
* A history of active TB greater than 3 years ago unless there is documentation that the prior anti-TB treatment was appropriate in duration and type.
* Therapy for latent TB which has not been completed as per local guidelines.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen L Jablonski Nowak, Ph.D., Principal Investigator — University of Colorado Denver Anschutz Medical Campus
Locations (2):
- United States (2):
  - University of Colorado Clinical and Translational Research Center (CTRC) Outpatient Clinic, Aurora, Colorado
  - Vanderbilt University Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rilonacept | Placebo
Started | 21 | 21
Completed | 18 | 19
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — dog bite | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rilonacept | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11) | 65 (11) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  White | 16 | 16 | 32
  Hispanic | 6 | 6 | 12
  African American | 5 | 5 | 10
Etiology of CKD [Number; unit: participants]
  Hypertension | 12 | 10 | 22
  Type II Diabetes | 10 | 9 | 19
  Type I DIabetes | 1 | 2 | 3
  Autosomal Dominant Polycystic Kidney Disease | 1 | 2 | 3
  Renal Cell Carcinoma | 0 | 3 | 3
  Focal Segmental Glomerulosclerosis | 1 | 0 | 1
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 38 (14) | 38 (12) | 38 (13)

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated Dilation (FMD)
Description: Change in FMD after 3 months of treatment with rilonacept will be compared to change in the placebo group.
Time Frame: 3 months after start of treatment
Measure: Mean (Standard Deviation); unit: change in percent flow-mediated dilation
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 18 | 19
change in percent flow-mediated dilation | 1.1 (3.2) | -0.9 (2.2)

2. Secondary Outcome: Change in Aortic Pulse-wave Velocity (aPWV)
Description: Change in aPWV after 3 months of treatment with rilonacept will be compared to change in the placebo group.
Time Frame: 3 months after start of treatment
Measure: Mean (Standard Deviation); unit: change in pulse-wave velocity (cm/sec)
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 18 | 19
change in pulse-wave velocity (cm/sec) | 12 (65) | 2 (71)

3. Secondary Outcome: Change in Contribution of Oxidative Stress to FMD
Description: FMD will be assessed following acute infusion of ascorbic acid compared to saline. The improvement in FMD with ascorbic acid reflects the degree of oxidative stress contributing to impairment in FMD.
Time Frame: 3 months after start of treatment
Population: sub-group from Denver site
Measure: Mean (Standard Deviation); unit: change in percent flow-mediated dilation
Groups:
- Rilonacept: Baseline: Change in flow-mediated dilation following an acute infusion of ascorbic acid (as compared to saline) in the rilonacept group at baseline.
- Rilonacept: End of Study: Change in flow-mediated dilation following an acute infusion of ascorbic acid (as compared to saline) in the rilonacept group at 12 weeks.
- Placebo: Baseline; Placebo: End of Study: Change in flow-mediated dilation following an acute infusion of ascorbic acid (as compared to saline) in the placebo group at baseline
Arm/Group | Rilonacept: Baseline | Rilonacept: End of Study | Placebo: Baseline | Placebo: End of Study
Number analyzed (Participants) | 10 | 7 | 13 | 10
change in percent flow-mediated dilation | 0.16 (2.52) | 0.51 (2.24) | -0.04 (1.96) | 0.69 (1.73)

4. Other Pre Specified Outcome: Change in High-sensitivity C-reactive Protein (hsCRP)
Description: Change in high-sensitivity C-reactive protein (hsCRP) after 3 months of rilonacept vs. placebo will be assessed as a circulating marker of inflammation.
Time Frame: 3 months after start of treatment
Measure: Median (Inter-Quartile Range); unit: change in c-reactive protein (mg/L)
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 16 | 19
change in c-reactive protein (mg/L) | -1.02 [-2.9 to 1.3] | 0.16 [-0.82 to 1.19]

5. Other Pre Specified Outcome: Change in Vascular Endothelial NADPH Oxidase Expression
Description: Vascular endothelial cells will be collected and assessed for changes in protein expression of NADPH oxidase after 3 months of treatment with rilonacept vs. placebo. Protein expression is calculated as a ratio of intensity of staining in the patient cells relative to human umbilical vein endothelial cell (HUVEC) control cells. The absolute change in this ratio between baseline and week 12 is reported below.
Time Frame: 3 months after start of treatment
Population: sub-group from Denver site
Measure: Mean (Standard Deviation); unit: absolute change in ratio
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 6 | 5
absolute change in ratio | -0.02 (0.03) | 0.01 (0.03)

ADVERSE EVENTS:
Arm/Group | Rilonacept | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 5/21 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rilonacept (N=21) | Placebo (N=21)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 | 1
Neck abscess/pyomyositis (Infections and infestations) | 1 | 0
upper respiratory infection (Infections and infestations) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No